CLINICAL TRIAL: NCT05634525
Title: Phase Ib Trial of the KRASG12C Inhibitor Adagrasib (MRTX849) in KRAS G12C Mutant Metastatic Pancreatic Cancer Patients
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Mirati Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0174; NCI-2022-10011 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2022-11-22; First posted 2022-12-02 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Metastatic Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — adagrasib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- MRTX849 (Adagrasib) (Experimental): Helps to control pancreatic cancer that has a KRAS G12 mutation.
  Interventions: Drug: MRTX849

INTERVENTIONS:
Drug: MRTX849 — Given By PO
  Other Names: Adagrasib

SUMMARY:
To learn if the investigational study drug, adagrasib (also called MRTX849), can help to control pancreatic cancer that has a KRAS G12 mutation. The safety and possible effects of adagrasib will also be studied.

DETAILED DESCRIPTION:
Primary Objectives:

To assess the preliminary antitumor activity of Adagrasib (MRTX849) monotherapy in metastatic pancreatic cancer patients with KRAS G12C mutation using Objective Response Rate (ORR) = Complete response (CR)+Partial response (PR) by RECIST 1.1 criteria1.

Secondary Objectives:

To evaluate the safety, tolerability and antitumor activity of Adagrasib (MRTX849) monotherapy in metastatic pancreatic cancer patients with KRASG12C mutation including median overall survival (OS), progression free survival (PFS), safety and adverse events (AEs).

Exploratory objectives:

Exploratory objectives include identiying the genomic and nongenomic mechanisms to responses and resistance and the specific immune cells involved with outcome.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following inclusion criteria to be eligible for enrollment into the study.

1. Histologically confirmed diagnosis of a pancreatic cancer with KRAS G12C mutation. Patients are eligible based on detection of KRAS G12C mutation in tumor tissue or plasma circulating tumor DNA (ctDNA) by any CLIA-certified lab assay.
2. Unresectable or metastatic disease.
3. Presence of tumor lesions to be evaluated per RECIST 1.1. Patients must have measurable or evaluable disease
4. Age ≥ 18 years old
5. Life expectancy of at least 3 months.
6. No more than one prior therapy. Prior systemic therapy (e.g., chemotherapy, immunotherapy or, investigational agent) and radiation therapy discontinued at least 2 weeks before first dose date.
7. Recovery from the adverse effects of prior therapy at the time of enrollment to ≤ Grade 1 (excluding alopecia and neuropathy).
8. Eastern Cooperative Oncology Group (ECOG) performance status in 0 to 2.
9. Laboratory values within the screening period:

   1. Absolute neutrophil count 1000/mm3 ( 1.0 x 109/L)
   2. Platelet count 75,000/mm3 ( 75 x 109/L)
   3. Hemoglobin ≥ 8 g/dL, in the absence of transfusions for at least 2 weeks
   4. Total bilirubin ≤2 x Upper Limit of Normal (ULN) (if associated with liver metastases or Gilbert's disease, ≤3 x ULN)
   5. Aspartate transaminase (AST) and alanine transaminase (ALT) ≤5 x ULN (if associated with liver metastases, ≤5 x ULN)
   6. Creatinine clearance ≥60 mL/min calculated using a validated prediction equation (e.g., Cockcroft-Gault, MDRD, or 24-hour urine CrCl) or serum creatinine 1.5XULN per institutional criterion.
10. Women of child-bearing potential (WOCBP) or men whose partner is a WOCBP agrees to use contraception while participating in this study, and for a period of 6 months following termination of study treatment.
11. Completed informed consent process, including signing IRB/EC-approved informed consent form.
12. Willing to comply with clinical trial instructions and requirements.
13. Patients who are biologically capable of having children and sexually active must agree to use an acceptable method of contraception for the duration of the treatment period and for at least 6 months after the last dose of study treatment. The local Investigator will counsel the patient on selection of contraception method and instruct the patient in its consistent and correct use. Examples of acceptable forms of contraception include:

    * Oral, inserted, injected or implanted hormonal methods of contraception, provided it has been used for an adequate period of time to ensure effectiveness.
    * Correctly placed copper containing intrauterine device (IUD).
    * Male condom or female condom used WITH a spermicide.
    * Male sterilization with confirmed absence of sperm in the post-vasectomy ejaculate.
    * Bilateral tubal ligation or bilateral salpingectomy. The local Investigator will instruct the patient to call immediately if the selected birth control method is discontinued or if pregnancy is known or suspected.

Note: Women are considered post-menopausal and/or not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g., age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least 6 months ago. In case of any ambiguity, the reproductive status of the woman should be confirmed by hormone level assessment.

Exclusion Criteria:

Patients presenting with any of the following will be excluded from the study:

1. Active brain metastases. Patients are eligible if brain metastases are adequately treated and patients are neurologically stable (except for residual signs or symptoms related to the central nervous system (CNS) treatment) for at least 2 weeks prior to enrollment without the use of corticosteroids or are on a stable or decreasing dose of ≤ 10 mg daily prednisone (or equivalent).
2. Carcinomatous meningitis
3. History of significant hemoptysis or hemorrhage with Hemoglobin dropped below 8 g/dL within 4 weeks of the first dose date.
4. Major surgery within 4 weeks of first dose date.
5. Inability to swallow oral medications.
6. Any of the following cardiac abnormalities:

   * Unstable angina pectoris or myocardial infarction within the previous 6 months
   * Congestive heart failure ≥NHYA Class 3 within the previous 6 months
   * LVEF<50%
   * QTcF > 480 milliseconds or medical or immediate family history of congenital Long QT Syndrome
7. Symptomatic or uncontrolled atrial fibrillation or other arrhythmia
8. History of stroke or transient ischemic attack within the previous 6 months.
9. Ongoing need for a medication with any of the following characteristics that cannont be switched to alternative treatment prior to study entry: known risk of QT prolongation or Torsades de Pointes; substrate of CYP3A with narrow therapeutic index; strong inducer of CYP3A and/or P-gp; strong inhibitor of BCRP; and proton pump inhibitors (see Table 17 and Table 18).
10. Second malignancy that either requires active concurrent systemic therapy or involves a lesion that may confound assessment of the pancreatic cancer under study.
11. Known active human immunodeficiency virus (HIV) or Hepatitis B or C. Note that the following are permitted:

    1. Patients treated for hepatitis C with no detectable viral load;
    2. Patients treated for HIV with no detectable viral load for at least 1 month prior to enrollment while on a stable regimen of agents that are not strong inhibitors of CYP3A4; and
    3. Patients with hepatitis B (HBV) receiving prophylaxis against reactivation of hepatitis B (either [HBsAg-positive with normal ALT and HBV DNA < 2,000 IU/mL or < 10,000 copies/mL] or [HBsAg-negative and anti-HBc-positive]).
12. Pregnancy. WOCBP must have a negative serum or urine pregnancy test documented within the screening period prior start of study drug.
13. Breast-feeding or planning to breast feed during the study or within 6 months after study treatment.
14. Any serious illness, uncontrolled inter-current illness, psychiatric illness, active or uncontrolled infection, or other medical history, including laboratory results, which, in the local Investigator's opinion, would be likely to interfere with the patient's participation in the study, or with the interpretation of the results.
15. Prior treatment with a therapy targeting KRAS G12C mutation is permitted

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-05-03 (Actual); Primary Completion 2025-07-21 (Actual); Study Completion 2025-07-21 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) | through study completion; an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Dan Zhao, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org